CLINICAL TRIAL: NCT00443846
Title: An Open-label, Randomised, Comparative, Multi-centre Study of the Immunogenicity and Safety of the Concomitant Use of a Live Pentavalent Rotavirus Vaccine (RotaTeq®) and a Meningococcal Group C Conjugate (MCC) Vaccine in Healthy Infants
Brief Title: RotaTeq® and Meningococcus C Vaccine in Healthy Infants (V260-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V260-016; S06-ROT-304 (Other: MCMVaccBV (SPMSD) Protocol Number); 2006-005445-11 (EudraCT Number)
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2017-09

CONDITIONS: Meningitis, Meningococcal; Rotavirus Infections
Keywords: Prevention of Gastroenteritis due to rotavirus infection. And prevention of Invasive disease caused by Neisseria meningitidis serogroup C.
MeSH Terms: conditions — Meningitis, Meningococcal; Rotavirus Infections | interventions — RotaTeq; Rotavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Concomitant Administration (Experimental): Participants received 2 concomitant doses of RotaTeq® and MCC vaccine at 10-11 weeks of age and 20-21 weeks of age and a third dose of RotaTeq® at 24-25 weeks of age (and 28 to 42 days after the vaccine administration at 20-21 weeks of age).
  Interventions: Biological: RotaTeq®; Biological: NeisVac-C®
- Group 2: Sequential Administration (Active Comparator): Participants received 3 doses of RotaTeq® at 6-7 weeks of age, 15-16 weeks of age, and 24-25 weeks of age (and 28 to 42 days after the MMC vaccine administered at 20-21 weeks of age), and MCC vaccine at 10-11 weeks of age and 20-21 weeks of age.
  Interventions: Biological: RotaTeq®; Biological: NeisVac-C®

INTERVENTIONS:
Biological: RotaTeq® — Rotavirus vaccine, live, oral, pentavalent, 2 mL solution for oral administration.
  Other Names: V260
Biological: NeisVac-C® — Meningiococcal Group C Polysaccharide Conjugate Vaccine Absorbed, 0.5 mL suspension for intramuscular injection.

SUMMARY:
Primary objective:

To check if RotaTeq® can be administered concomitantly with meningococcal Group C vaccine without impairing the efficacy of MCC vaccine. The hypothesis tested is that the seroprotection rate for MMC at 28 days after the second MCC vaccination with concomitant administration of RotaTeq® is non-inferior to that without non-concomitant (sequential) administration of RotaTeq®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, aged from 6 weeks through full 7 weeks,
* Consent form signed by at least one parent or by the legal representative properly informed about the study,
* Parent(s) / legal representative able to understand the protocol requirements and to fill in the Diary Card.

Exclusion Criteria:

* History of congenital abdominal disorders, congenital malformation of the gastrointestinal tract that could predispose to intussusception, or abdominal surgery,
* Congenital fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency,
* Known or suspected impairment of immunological function,
* Known hypersensitivity to any component of RotaTeq® (e.g. sucrose) or of NeisVac-C® (including tetanus toxoid),
* Prior administration of any rotavirus vaccine,
* Prior administration of any vaccine within the 28 days prior to randomisation,
* Fever (rectal temperature ≥38.1°C) and/or acute diarrhoea and/or vomiting at randomisation,
* History of known prior rotavirus gastroenteritis, chronic diarrhoea, or failure to thrive,
* Any severe thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection,
* Clinical evidence of active gastrointestinal illness,
* Receipt of intramuscular, oral, or intravenous corticosteroid treatment within the 14 days prior to randomisation. Note: Infants on inhaled and/or topical steroids may participate in the study,
* Infants residing in a household with an immunocompromised person,
* Prior receipt of a blood transfusion or blood products, including immunoglobulins.

Ages: 42 Days to 55 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 247 (Actual)
Dates: Start 2007-02-13 (Actual); Primary Completion 2007-09-04 (Actual); Study Completion 2007-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Vesikari T, Karvonen A, Borrow R, Kitchin N, Baudin M, Thomas S, Fiquet A. Results from a randomized clinical trial of coadministration of RotaTeq, a pentavalent rotavirus vaccine, and NeisVac-C, a meningococcal serogroup C conjugate vaccine. Clin Vaccine Immunol. 2011 May;18(5):878-84. doi: 10.1128/CVI.00437-10. Epub 2011 Mar 9. PMID 21389149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 249 participants were screened and 247 were randomized.
Period: Overall Study
Arm/Group | Group 1: Concomitant Administration | Group 2: Sequential Administration
Started | 124 | 123
Vaccinated | 116 | 123
Completed | 113 | 117
Not Completed | 11 | 6
Not completed — Withdrawn due to intercurrent disease | 1 | 0
Not completed — Not vaccinated, no blood sample drawn | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Personal reason | 8 | 3
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Concomitant Administration | Group 2: Sequential Administration | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.1 (0.5) | 7.2 (0.6) | 7.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 55 | 105
  Male | 74 | 68 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroresponse for Meningiococcal Group C Serotype
Description: Antibody seroprotection to meningiococcal Group C serotype was measured by serum bactericidal antibody with rabbit complement (sRBA). The criterion for seroresponse was an sRBA titer >=1:8.
Time Frame: 28 days after the second dose of MCC vaccine (approximately 20 weeks)
Population: The population analyzed was randomized participants excluding those with protocol violations that may have interfered with the immunogenicity evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Concomitant Administration | Group 2: Sequential Administration
Number analyzed (Participants) | 104 | 106
Percentage of participants | 100 [96.5 to 100] | 100 [96.6 to 100]
Statistical Analysis 1: Comparison: Group 1: Concomitant Administration vs Group 2: Sequential Administration; Analysis of non-inferiority was based on the Miettinen and Nurminen method; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower bound of the 95% confidence interval of the difference (Group 1 - Group 2) in seroprotection rate was greater than -10%; Difference (Group 1 - Group 2) = 0, 95% CI 2-sided [-3.7 to 3.7]

ADVERSE EVENTS:
Time Frame: Serious and other adverse events: up to 13 days after any vaccination visit; solicited diarrhea, vomiting, and temperature: up to 6 days after any vaccination visit; deaths and vaccine- or procedure-related serious adverse events: up to 27 weeks.
Description: The population at risk was all vaccinated participants. One participant in Group 2 was excluded because they were lost to follow-up after receiving only the first dose of RotaTeq®.
Arm/Group | Group 1: Concomitant Administration | Group 2: Sequential Administration
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/122
Other Adverse Events (participants affected / at risk) | 98/116 | 105/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Concomitant Administration (N=116) | Group 2: Sequential Administration (N=122)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Concomitant Administration (N=116) | Group 2: Sequential Administration (N=122)
Conjunctivitis (Eye disorders) | 4 (5) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8) | 16 (21)
Diarrhoea (Gastrointestinal disorders) | 38 (52) | 48 (73)
Flatulence (Gastrointestinal disorders) | 9 (11) | 21 (26)
Regurgitation of food (Gastrointestinal disorders) | 6 (7) | 13 (15)
Teething (Gastrointestinal disorders) | 7 (8) | 2 (2)
Vomiting (Gastrointestinal disorders) | 30 (36) | 27 (40)
Injection-site erythema (General disorders) | 26 (30) | 23 (24)
Injection-site induration (General disorders) | 4 (5) | 7 (8)
Injection-site pain (General disorders) | 10 (11) | 6 (6)
Injection-site swelling (General disorders) | 6 (7) | 10 (11)
Irritability (General disorders) | 59 (76) | 51 (79)
Pyrexia (General disorders) | 32 (38) | 34 (36)
Rhinitis (Infections and infestations) | 13 (14) | 21 (26)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 10 (11)
Somnolence (Nervous system disorders) | 8 (10) | 9 (10)
Crying (Psychiatric disorders) | 12 (16) | 25 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.